CLINICAL TRIAL: NCT02548468
Title: A Two-Step Approach to Reduced Intensity Allogeneic Hematopoietic Stem Cell Transplantation for Advanced Cutaneous T Cell Lymphoma
Brief Title: Reduced Intensity Conditioning Before Partially Matched Donor Stem Cell Transplant in Treating Patients With Advanced Cutaneous T Cell Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15D.237; JT 6812 (Other: JeffTrial Number)
Record Dates: First submitted 2015-09-08; First posted 2015-09-14 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Cutaneous T-Cell Non-Hodgkin Lymphoma; Recurrent Mycosis Fungoides and Sezary Syndrome; Stage IIB Mycosis Fungoides and Sezary Syndrome; Stage IIIA Mycosis Fungoides and Sezary Syndrome; Stage IIIB Mycosis Fungoides and Sezary Syndrome; Stage IVA Mycosis Fungoides and Sezary Syndrome; Stage IVB Mycosis Fungoides and Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — fludarabine; fludarabine phosphate; Whole-Body Irradiation; Cyclophosphamide; Peripheral Blood Stem Cell Transplantation; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Reduced Intensity Conditioning, DLI, PBSCT (Experimental): REDUCED INTENSITY CONDITIONING: Patients receive fludarabine phosphate IV over 30 minutes on days -11 to -8 and undergo total body irradiation BID on day -7. Patients also receive donor CD3+ enriched T lymphocyte infusion on day -6 and high-dose cyclophosphamide IV over 2 hours on days -3 to -2.
  TRANSPLANT: Patients undergo allogeneic PBSCT on day 0.
  GVHD PROPHYLAXIS: Beginning on day -1, patients receive tacrolimus IV with taper (drug wean) by day 60 and mycophenolate mofetil IV BID on days -1 to 28 in the absence of GVHD.
  Interventions: Drug: Fludarabine; Radiation: Total-Body Irradiation; Biological: T Cell-Depleted Donor Lymphocyte Infusion; Drug: Cyclophosphamide; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Mycophenolate mofetil; Drug: Tacrolimus

INTERVENTIONS:
Drug: Fludarabine — Given IV
  Other Names: Fludarabine phosphate; Fludara
Radiation: Total-Body Irradiation — Undergo TBI
Biological: T Cell-Depleted Donor Lymphocyte Infusion — Undergo donor CD3+ enriched T lymphocyte infusion
Drug: Cyclophosphamide — Given IV
  Other Names: Endoxan; Cytoxan; Neosar; Procytox; Revimmune; Cycloblastin; Cytophosphane; CP
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic HSC transplant
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo allogeneic PBSCT
Drug: Mycophenolate mofetil — Given IV
  Other Names: MMF
Drug: Tacrolimus — Given IV
  Other Names: FK-506; Fujimycin; Prograf; Advagraf; Protopic

SUMMARY:
This phase I trial studies the side effects and the best dose of donor lymphocyte infusion when given together with reduced intensity conditioning regimen before partially matched donor stem cell transplant in treating patients with stage IIB-IV mycosis fungoides or Sezary syndrome. Giving chemotherapy and low-dose total-body irradiation followed by high-dose cyclophosphamide before a donor peripheral blood stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft-versus-host disease). Removing the T-cells from the donor cells and giving them before transplant may stop this from happening. Additionally, giving tacrolimus and mycophenolate mofetil before and after transplant may also stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTVES:

I. To evaluate regimen related toxicity, engraftment and graft versus host disease (GVHD) in the first 100 days with new reduced intensity haploidentical regimen protocol, including fludarabine (fludarabine phosphate), low dose total body irradiation, and cyclophosphamide.

II. To determine an effective donor lymphocyte infusion (DLI) dose that provides successful engraftment without causing GVHD.

SECONDARY OBJECTIVES:

I. To assess myeloid and lymphoid engraftment rates of patients undergoing treatment on this regimen.

II. To determine the incidence and severity of GVHD in patients undergoing treatment on this regimen using a combination of tacrolimus and mycophenolate mofetil (MMF) as GVHD prophylaxis.

III. To examine progression free survival and overall survival in patients with cytotoxic T-cell lymphoma (CTCL) undergoing treatment on this regimen.

IV. To assess the pace of lymphoid recovery in this patient population.

OUTLINE: This is a phase I, dose-escalation study of DLI.

REDUCED INTENSITY CONDITIONING: Patients receive fludarabine phosphate intravenously (IV) over 30 minutes on days -11 to -8 and undergo total body irradiation twice daily (BID) on day -7. Patients also receive donor cluster of differentiation (CD)3+ enriched T lymphocyte infusion on day -6 and high-dose cyclophosphamide IV over 2 hours on days -3 to -2.

TRANSPLANT: Patients undergo allogeneic peripheral blood stem cell transplant (PBSCT) on day 0.

GVHD PROPHYLAXIS: Beginning on day -1, patients receive tacrolimus IV with taper (drug wean) by day 60 and mycophenolate mofetil IV BID on days -1 to 28 in the absence of GVHD.

After completion of treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IIB-IV mycosis fungoides and sezary syndrome who have failed at least one standard systemic therapy or are not candidates for standard therapy.
2. Patient should have a responsive skin disease including complete remission (CR) and partial remission (PR) (close to CR; 75%-99% clearance of skin disease from baseline without new tumors (T3) in patients with T1, T2 or T4 only skin disease) and should not have visceral organ or lymph node involvement prior to transplantation.
3. Patients must have a related donor who is a two or more allele mismatch at the HLA-A; B; C; DR and DQ loci. Patients who have sibling donors with a one antigen mismatch due to recombination will not be enrolled in this protocol.
4. Patients must have adequate organ function:

   * Left Ventricular Ejection Fraction (LVEF) of >50%
   * Carbon Monoxide Diffusing Capacity (DLCO) >50% of predicted corrected for hemoglobin
   * Adequate liver function as defined by a serum bilirubin <2.0 (unless hemolysis or Gilbert disease), Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) < 2.5 X upper limit of normal
   * Creatinine clearance of > 60 ml/min
5. Performance status > 80% (Karnofsky)
6. Hematopoietic Cell Transplantation Specific Comorbidity Index (HCT-CI) <5 for age < 65, HCT-CI <4 for age >65
7. Patients must be willing to use contraception if they have childbearing potential
8. Able to give informed consent, or their legally authorized representative can give informed consent.

Exclusion Criteria:

1. Performance status of < 80% (Karnofsky)
2. HIV positive
3. Active involvement of the central nervous system with malignancy
4. Psychiatric disorder that would preclude patients from signing an informed consent
5. Pregnancy, or unwillingness to use contraception if they are have childbearing potential.
6. Patients with life expectancy of < 6 months for reasons other than their underlying hematologic/oncologic disorder or complications there from.
7. Patients who have received alemtuzumab within 8 weeks of transplant admission, or who have recently received horse or rabbit anti-thymocyte globulin (ATG) and have ATG levels of > 2 μgm/ml.
8. Patients who cannot receive cyclophosphamide
9. Patients with evidence of another malignancy (exclusive of a skin cancer that requires only local treatment);

   * Patients with prior malignancies diagnosed> 5 years ago without evidence of disease are eligible.
   * Patients with prior malignancy treated < 5 years ago but have a life expectancy of > 5 years for that malignancy are eligible.
10. Uncontrolled active infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11-20 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-03-16 (Actual)

PRIMARY OUTCOMES:
Rate of regimen-related toxicities | Up to 100 days post-transplant
  Estimate of dose-specific rates of toxicity will be presented with corresponding confidence intervals using the exact method. The method of Atkinson and Brown will be used for any rate related to definition of dose limiting toxicity, due to two-stage sampling.
Rate for hematopoietic engraftment | Up to 100 days post-transplant
  Estimate of dose-specific rate for engraftment will be presented with corresponding confidence intervals using the exact method. The method of Atkinson and Brown will be used for any rate related to definition of dose limiting toxicity, due to two-stage sampling.
Rate for immune reconstitution | Up to 100 days post-transplant
  Estimate of dose-specific rate for immune reconstitution will be presented with corresponding confidence intervals using the exact method. The method of Atkinson and Brown will be used for any rate related to definition of dose limiting toxicity, due to two-stage sampling.
Incidence of GVHD | Up to 100 days post-transplant
Maximum tolerated dose of DLI, determined according to dose limiting toxicities | day -4

SECONDARY OUTCOMES:
Myeloid engraftment rate | Up to 6 months post-transplant
Lymphoid engraftment rate | Up to 6 months post-transplant
Incidence of GVHD using tacrolimus and mycophenolate mofetil prophylaxis | Up to 6 months post-transplant
Progression free survival | Up to 6 months post-transplant
  Progression free survival will be estimated by the Kaplan-Meier method.
Overall survival (OS) | Up to 6 months post-transplant
  OS will be estimated by the Kaplan-Meier method.
Rate of lymphoid recovery | Up to 6 months post-transplant
Incidence of adverse events | Up to 6 months
  All estimates of dose-specific rates (e.g., toxicity) will be presented with corresponding confidence intervals using the exact method. The method of Atkinson and Brown will be used for any rate related to definition of dose limiting toxicity, due to two-stage sampling.

CONTACTS AND LOCATIONS:
Overall Officials: S. Onder Alpdogan, MD, Principal Investigator — Thomas Jefferson University

REFERENCES:
- See also: Sidney Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Jefferson University Hospitals — http://hospitals.jefferson.edu/